CLINICAL TRIAL: NCT00622661
Title: A Feeding Study to Examine the Effect of Glycemic Load and Obesity on Cancer Biomarkers
Brief Title: Carbohydrates and Related Biomarkers
Acronym: CARB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Marian Neuhouser, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PHS 2059.00; NIH/NCI U54 CA 116847; IR 6105
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Healthy; Overweight
Keywords: Glycemic response; Glycemic index; Obesity; Carbohydrates; Insulin; Blood glucose
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Normal weight
  Interventions: Other: Low Glycemic Load Diet; Other: High Glycemic Load Diet
- 2 (Other): Overweight
  Interventions: Other: Low Glycemic Load Diet; Other: High Glycemic Load Diet

INTERVENTIONS:
Other: Low Glycemic Load Diet — consume both high and low glycemic load diets for 28 days each
Other: High Glycemic Load Diet — consume both high and low glycemic load diets for 28 days each

SUMMARY:
This study is designed to investigate associations of low- and high-glycemic load diets with biomarkers of hyperglycemia, hyperinsulinemia and inflammation, potential biomarkers for cancer risk.

DETAILED DESCRIPTION:
This is a randomized, crossover feeding study conducted in normal weight and overweight individuals. Participants will be given all their food to eat and drink (except water) for two 28-day feeding periods (a total of 56 days). The diets will be carefully controlled and energy intake will be regulated to maintain weight stability for each participant. The two feeding periods will be separated by a 28 day "washout" period when participants will eat their own food. Dinner will be eaten at the Hutchinson Center Monday through Friday. Each evening, breakfast, lunch and snacks will be brought home for the next day. On Friday evenings all the food will be taken home for the weekend.

Samples of blood will be collected after an overnight fast at the beginning and the end of each feeding period. All urine will be collected for 24 hours at the end of each feeding period. A number of questionnaires will also be completed during each diet period. A small stool sample will be collected in your own home, before the first feeding period, and once during each feeding period. The stool sample collection is optional. One can decide not to provide a stool sample and still participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and female subjects
2. Between the ages of 18 to 45
3. BMI between 18.5 kg/m2 to 24. 9 kg/m2 (normal weight) and between 28.0 kg/m2 to 39.9 kg/m2 (overweight)
4. Willingness to refrain from alcohol during the study
5. Able to come to the FHCRC in Seattle every weekday night for dinner

Exclusion Criteria:

1. Younger than 18 years of age or older than 45 years of age.
2. Do not fit into one of the study weight groups (normal weight and overweight): BMI < 18.5 kg/m2 or > 40.0 kg/m2, and between 25.0 kg/m2and 27.9 kg/m2
3. Have diseases that are treated by diet and/or medications including but not limited to diabetes, kidney disease, heart disease
4. Taking prescription medications every day (this includes women taking birth-control pills, shots, patch or IUD with hormones)
5. Diagnosed with or treated for cancer within the previous five years (except those with a diagnosis and/or treatment of non-melanomatous skin cancer are eligible)
6. Currently pregnant or breastfeeding or planning a pregnancy in the next 3 months.
7. Using any tobacco products on a daily basis (cigarettes, pipes, cigars, chewing tobacco).
8. Using recreational drugs
9. Drinking the following amount of alcohol almost every day: 2 or more cans/bottles of beer OR 2 or more glasses of wine OR 3 or more ounces of hard liquor.
10. Inability (e.g., food allergy or intolerances) or unwillingness to consume the foods that are part of the feeding study diet.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2006-06; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoints of the study will be a set of inter-related biomarkers for hyperglycemia, hyperinsulinemia and inflammation, potential biomarkers for cancer risk. | two 4-week feeding periods (56 days total)

SECONDARY OUTCOMES:
Questionnaires will generate data on how these diets may influence mood or depression, sleep habits, and measures of appetite and satiety. | two 4-week feeding periods (56 days)

CONTACTS AND LOCATIONS:
Overall Officials: Marian Neuhouser, RD, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Hullar MA, Kahsai O, Curtis KR, Navarro SL, Zhang Y, Randolph TW, Levy L, Shojaie A, Kratz M, Neuhouser ML, Lampe PD, Raftery D, Lampe JW. Metabolic plasticity of the gut microbiome in response to diets differing in glycemic load in a randomized, crossover, controlled feeding study. Am J Clin Nutr. 2025 Sep;122(3):780-792. doi: 10.1016/j.ajcnut.2025.06.026. Epub 2025 Jul 5. PMID 40619005
- [Derived] Dibay Moghadam S, Navarro SL, Shojaie A, Randolph TW, Bettcher LF, Le CB, Hullar MA, Kratz M, Neuhouser ML, Lampe PD, Raftery D, Lampe JW. Plasma lipidomic profiles after a low and high glycemic load dietary pattern in a randomized controlled crossover feeding study. Metabolomics. 2020 Nov 20;16(12):121. doi: 10.1007/s11306-020-01746-3. PMID 33219392
- [Derived] Navarro SL, Tarkhan A, Shojaie A, Randolph TW, Gu H, Djukovic D, Osterbauer KJ, Hullar MA, Kratz M, Neuhouser ML, Lampe PD, Raftery D, Lampe JW. Plasma metabolomics profiles suggest beneficial effects of a low-glycemic load dietary pattern on inflammation and energy metabolism. Am J Clin Nutr. 2019 Oct 1;110(4):984-992. doi: 10.1093/ajcn/nqz169. PMID 31432072
- [Derived] Ginos BNR, Navarro SL, Schwarz Y, Gu H, Wang D, Randolph TW, Shojaie A, Hullar MAJ, Lampe PD, Kratz M, Neuhouser ML, Raftery D, Lampe JW. Circulating bile acids in healthy adults respond differently to a dietary pattern characterized by whole grains, legumes and fruits and vegetables compared to a diet high in refined grains and added sugars: A randomized, controlled, crossover feeding study. Metabolism. 2018 Jun;83:197-204. doi: 10.1016/j.metabol.2018.02.006. Epub 2018 Feb 17. PMID 29458053
- [Derived] Breymeyer KL, Lampe JW, McGregor BA, Neuhouser ML. Subjective mood and energy levels of healthy weight and overweight/obese healthy adults on high-and low-glycemic load experimental diets. Appetite. 2016 Dec 1;107:253-259. doi: 10.1016/j.appet.2016.08.008. Epub 2016 Aug 6. PMID 27507131
- [Derived] Barton S, Navarro SL, Buas MF, Schwarz Y, Gu H, Djukovic D, Raftery D, Kratz M, Neuhouser ML, Lampe JW. Targeted plasma metabolome response to variations in dietary glycemic load in a randomized, controlled, crossover feeding trial in healthy adults. Food Funct. 2015 Sep;6(9):2949-56. doi: 10.1039/c5fo00287g. PMID 26165375
- [Derived] Runchey SS, Pollak MN, Valsta LM, Coronado GD, Schwarz Y, Breymeyer KL, Wang C, Wang CY, Lampe JW, Neuhouser ML. Glycemic load effect on fasting and post-prandial serum glucose, insulin, IGF-1 and IGFBP-3 in a randomized, controlled feeding study. Eur J Clin Nutr. 2012 Oct;66(10):1146-52. doi: 10.1038/ejcn.2012.107. Epub 2012 Aug 15. PMID 22892437
- [Derived] Chang KT, Lampe JW, Schwarz Y, Breymeyer KL, Noar KA, Song X, Neuhouser ML. Low glycemic load experimental diet more satiating than high glycemic load diet. Nutr Cancer. 2012;64(5):666-73. doi: 10.1080/01635581.2012.676143. Epub 2012 May 7. PMID 22564018
- [Derived] Neuhouser ML, Schwarz Y, Wang C, Breymeyer K, Coronado G, Wang CY, Noar K, Song X, Lampe JW. A low-glycemic load diet reduces serum C-reactive protein and modestly increases adiponectin in overweight and obese adults. J Nutr. 2012 Feb;142(2):369-74. doi: 10.3945/jn.111.149807. Epub 2011 Dec 21. PMID 22190020